CLINICAL TRIAL: NCT06406517
Title: Comparative Effectiveness of Gadopiclenol for Evaluation of Adult Congenital Heart Anatomy and Hemodynamics
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Bracco Imaging S.p.A. (Industry)
Responsible Party: Principal Investigator, Albert Hsiao, Professor in Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: IRB #809813
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — gadopiclenol; gadobenic acid

STUDY DESIGN:
Intervention Model Description: This will be a prospective, single center, parallel group, double-blinded, randomized clinical trial. The study will be conducted at UC San Diego MRI suites. Study participants will be randomized into one of four study arms prior to their MRI: Gadopiclenol 0.075 mmol/kg, gadopiclenol 0.10 mmol/kg, gadopiclenol 0.15 mmol/kg, gadobenate dimeglumine 0.15 mmol/kg (standard of care).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study investigator/postdoctoral researcher/research coordinator will randomize participants into a study arm based on the day the participant is scheduled to receive their MRI. Participants will not be told which study arm they are being randomized into. MRI techs will be told which arm patients are randomized in to so that the correct IV contrast drug and dose will be administered. All MRIs will be read by cardiac radiologists, who will also not be told which study arm a participant was in. The master list of randomized participants will be maintained by the study investigator/postdoctoral researcher/research coordinator.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Gadobenate dimeglumine 0.15 mmol/kg (standard of care) (Active Comparator)
  Interventions: Drug: Gadobenate dimeglumine
- Gadopiclenol 0.075 mmol/kg (Experimental)
  Interventions: Drug: Gadopiclenol
- Gadopiclenol 0.10 mmol/kg (Experimental)
  Interventions: Drug: Gadopiclenol
- Gadopiclenol 0.15 mmol/kg (Experimental)
  Interventions: Drug: Gadopiclenol

INTERVENTIONS:
Drug: Gadopiclenol — Gadopiclenol is an FDA-approved gadolinium-based contrast agent (GBCA) for neurological and abdominal contrast-enhanced MRI. Participants will receive this contrast agent at one of three different doses prior to undergoing a congenital heart cardiac MRI/MRA. This contrast agent will be compared to gadobenate dimeglumine, the standard-of-care.
  Other Names: Vueway
  Arms: Gadopiclenol 0.075 mmol/kg; Gadopiclenol 0.10 mmol/kg; Gadopiclenol 0.15 mmol/kg
Drug: Gadobenate dimeglumine — Gadobenate dimeglumine is an FDA-approved GBCA that is used in standard clinical practice at UCSD for contrast-enhanced MRI/MRA studies, including cardiac MRI/MRA. This contrast agent is the standard of care to which gadopiclenol will be compared.
  Other Names: Multihance
  Arms: Gadobenate dimeglumine 0.15 mmol/kg (standard of care)

SUMMARY:
The goal of this clinical trial is to learn how well and at what doses gadopiclenol, a new intravenous (IV) contrast agent used for MRI, works to produce high-quality MRI images of the heart, in patients with a history of congenital heart disease, when compared to gadobenate dimeglumine, the IV contrast agent that is normally used at our institution for heart (cardiac) MRI. The main questions it aims to answer are:

* Does using gadopiclenol result in similar or superior image quality, similar signal-to-noise ratio (SNR), and similar flow measurements with 4-dimensional (4D) flow cardiac MRI when compared to gadobenate dimeglumine?
* At what dose(s) does gadopiclenol result in similar image quality (using the above metrics) for cardiac MRI when compared to gadobenate dimeglumine?

Researchers will compare cardiac MRI images obtained after administration of gadopiclenol to cardiac MRI images obtained after administration of gadobenate dimeglumine (called the standard of care treatment) to see if the images are of similar or superior quality.

Participants will:

* Be randomized to receive either gadopiclenol at one of three different doses or gadobenate dimeglumine before their congenital heart cardiac MRI
* Undergo their congenital heart cardiac MRI as they would during the course of normal clinical care.

DETAILED DESCRIPTION:
At the University of California San Diego (UCSD), we have developed a premier advanced clinical cardiovascular imaging program, which is a critical component of our Adult Congenital Heart Association (ACHA)-accredited adult congenital heart program. Central to these programs is 4D Flow MRI, which enables hemodynamic assessment of patients with repaired and unrepaired congenital heart disease. Adults with congenital heart disease require routine MRI for surveillance and management of complications of disease and repairs, and 4D Flow allows us to reliably perform these exams efficiently and accurately. Multiple works by our group, and confirmed by others, have highlighted the value of 4D Flow MRI for evaluating this patient population, and for vascular imaging applications beyond the heart.

Gadopiclenol is a recently FDA-approved intravenous, extracellular gadolinium contrast agent indicated for use in MRI. Though it has been shown to be effective in detection of central nervous system (CNS) lesions and of lesions outside the CNS, its performance in cardiovascular imaging is unknown, particularly in cardiac MRI performed for evaluation of adult congenital heart disease. We therefore seek to evaluate whether use of gadopiclenol results in superior image quality compared to, and therefore may be used in place of, gadobenate dimeglumine, our current standard of care in 4D Flow MRI and MR Angiography (MRA).

In our current clinical practice, like many others, gadobenate dimeglumine at 0.3 mL/kg (0.15 mmol/kg) is our standard of care for vascular enhancement and cardiac MRI, favored due to its long blood pool residence time, which parallels the longer acquisition time for 4D Flow MRI (~10 minutes), and its strong T1 shortening properties. Gadopiclenol, with its stronger T1 shortening properties and similar pharmacokinetics, may achieve similar effects but as a macrocyclic agent is a more stable gadolinium agent, and theoretically may have a better retention profile than older linear agents due to its lower approved dose. We therefore seek to determine whether gadopiclenol may be used in place of gadobenate dimeglumine for contrast-enhanced 4D Flow MRI and MRA. Since the optimal dose of gadopiclenol for this purpose is unknown, we will assess the relative performance of gadopiclenol across a dose range.

Standard dosing for gadopiclenol for CNS and abdominal imaging in adult and pediatric patients is 0.05 mmol/kg actual body weight (equivalent to 0.1 mL/kg). However, its safety has been evaluated at doses ranging from 0.025 mmol/kg to 0.3 mmol/kg. We therefore plan to assess the signal to noise ratio and image quality of patients undergoing cardiac MRI using gadopiclenol at three doses (0.075 mmol/kg, 0.10 mmol/kg, 0.15 mmol/kg) against our standard of care (gadobenate dimeglumine at 0.3 mL/kg (0.15 mmol/kg)). We hypothesize that gadopiclenol at each dose will be non-inferior to gadobenate dimeglumine, achieving similar qualitative image quality, similar SNR, and similar standard deviation amongst flow measurements with 4D Flow MRI. There is a strong possibility that gadopiclenol at an equimolar gadolinium dose to gadobenate dimeglumine will provide superior qualitative image quality and superior SNR in contrast-enhanced MRA and reduce standard deviation amongst flow measurements with 4D Flow MRI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* History of congenital heart disease and scheduled to undergo standard of care cardiac MRI and chest MRA as part of routine clinical care
* English is patient's primary spoken language

Exclusion Criteria:

* Pediatric patients
* Pregnant patients
* Patients with ongoing acute kidney injury (AKI) or severe, chronic kidney disease (GFR < 30 mL/min/1.73m2)
* History of hypersensitivity reaction to gadolinium based contrast agent
* English is not the patient's primary spoken language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Image Quality | Image Quality will be assessed on a rolling basis during the study by all radiologists and will be completed within one month of the conclusion of enrollment.
  Images will be qualitatively scored by three attending radiologists for quality of contrast enhancement on a 5-point likert Scale
Signal-to-Noise Ratio (SNR) | SNR will be assessed on a rolling basis during the study by the study team and will be completed within one month of the conclusion of enrollment.
  Signal-to-noise will be measured from the blood pool in the aorta and main pulmonary artery and compared against myocardial signal for contrast-to-background calculations in contrast-enhanced MRA and 4D Flow signal images. This ca be readily performed by placing a region of interest (ROI) within the vessel of interest and calculating the standard deviation of signal intensities relative to mean signal intensity.
Standard Deviation of Volumetric Flow Measurements | Standard deviation of flow measurements will be assessed on a rolling basis during the study by all attending radiologists and will be completed within one month after the conclusion of enrollment.
  We will measure standard deviation of volumetric flow measurements from the aorta and main pulmonary artery from ROIs that are typically used in our clinical routine to measure systemic and pulmonary blood flow. The standard error in these measurements will be compared between each of the four randomized conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Hsiao, MD/PhD, Principal Investigator — Department of Radiology, UC San Diego
Locations (1):
- University of California San Diego Health, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobs K, Hahn L, Horowitz M, Kligerman S, Vasanawala S, Hsiao A. Hemodynamic Assessment of Structural Heart Disease Using 4D Flow MRI: How We Do It. AJR Am J Roentgenol. 2021 Dec;217(6):1322-1332. doi: 10.2214/AJR.21.25978. Epub 2021 Jun 2. PMID 34076463
- [Background] Kebebew E, Tresler PA, Siperstein AE, Duh QY, Clark OH. Normal thyroid pathology in patients undergoing thyroidectomy for finding a RETgene germline mutation: a report of three cases and review of the literature. Thyroid. 1999 Feb;9(2):127-31. doi: 10.1089/thy.1999.9.127. PMID 10090311
- [Background] Hsiao A, Alley MT, Massaband P, Herfkens RJ, Chan FP, Vasanawala SS. Improved cardiovascular flow quantification with time-resolved volumetric phase-contrast MRI. Pediatr Radiol. 2011 Jun;41(6):711-20. doi: 10.1007/s00247-010-1932-z. Epub 2011 Jan 11. PMID 21221566